CLINICAL TRIAL: NCT05687279
Title: Phase II, Randomized, Observer-blind, Placebo-controlled, Multi-center Study of a Live Attenuated Respiratory Syncytial Virus Vaccine to Assess the Vaccine Virus' Transmissibility in Household or Daycare Center Settings, Shedding, and Genetic Stability, and to Describe the Immunogenicity and Safety of the Vaccine in Infants and Toddlers 6 to < 24 Months of Age in Puerto Rico (USA)
Brief Title: Study on a Live-attenuated Respiratory Syncytial Virus Vaccine for Assessment of Safety, Transmissibility, and Genetic Stability of the Vaccine Virus Among Close Contacts in Infants and Toddlers 6 to < 24 Months of Age in Puerto Rico (USA)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAD00014; U1111-1278-3910 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind:
  * Blinding for vaccine group assignment: participants, parents or legally acceptable representative (LAR), outcome assessors, investigators, laboratory personnel, Sponsor study staff
  * No blinding for study staff who prepare and administer the study interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVt Vaccine Group (Experimental): 2 intranasal administrations (56 days apart) of the RSVt vaccine at D01 and D57
  Interventions: Biological: RSVt Vaccine
- Control Group (Placebo Comparator): 2 intranasal administrations (56 days apart) of the placebo at D01 and D57
  Interventions: Other: Control Group

INTERVENTIONS:
Biological: RSVt Vaccine — Pharmaceutical Form: Suspension of virus in a nasal spray Route of Administration: Intranasal
  Arms: RSVt Vaccine Group
Other: Control Group — Pharmaceutical Form: Suspension of virus in a nasal spray Route of Administration: Intranasal
  Arms: Control Group

SUMMARY:
The primary purpose of the study is to assess the shedding, transmission, and genetic stability of the live-attenuated RSVt vaccine after each intranasal vaccination (56 days apart) in infants and toddlers 6 to < 24 months of age.

DETAILED DESCRIPTION:
The duration of each participant's participation is up to 8 months, including the 6 months safety follow-up phone call after the second study intervention administration for the pediatric participants The treatment administration for the pediatric participants will be on D01 and D57 (1 intranasal administration each).

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to < 24 months on the day of inclusion (from the day of the 6 months after birth to the day before the 2nd birthday)
* Participants who are healthy as determined by medical evaluation including medical history.
* Born at full term of pregnancy (≥ 37 weeks) or born after a gestation period of 27 through 36 weeks and medically stable as assessed by the investigator, based on the following definition: "Medically stable" refers to the condition of premature infants who do not require significant medical support or ongoing management for debilitating disease and who have demonstrated a clinical course of sustained recovery by the time they receive the first dose of study intervention
* Attends a daycare facility at least 3 days per week and 4 hours per day at which the participant would be in a contact group/playroom of at least one other child 6 to < 24 months of age who will participate in this study or is a member of a household, which includes at least one other child 6 to < 24 months of age who will participate in this study

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Any acute febrile illness in the past 48 hours that according to investigator judgment is significant enough to interfere with successful inoculation on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Probable or confirmed ongoing case of COVID-19 at the time of enrollment
* Member of a household that contains an immunocompromised individual, including, but not limited to:

  * a person who is HIV infected
  * a person who has received chemotherapy within the 12 months prior to study enrollment
  * a person who has received (within the past 6 months) or is receiving (at the time of enrollment) immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Member of a household that includes, or will include, an infant who is less than 6 months of age at the time of enrollment
* Attends a daycare facility and shares a daycare room with infants less than 6 months of age, and parent/legally acceptable representative is unable or unwilling to suspend attendance at the daycare facility for 28 days following study intervention administration
* Any need of supplemental oxygen therapy in a home or hospital setting at the time of enrollment.
* Participant's mother previous receipt or planned administration of an investigational RSV vaccine or any monoclonal antibody (such as Infliximab) during pregnancy and/or breastfeeding.
* Receipt or planned receipt of any of the following vaccines prior to or after the first study intervention administration:

  * any influenza vaccine within 7 days prior to and after, or any COVID-19 or inactivated vaccine or live-attenuated rotavirus vaccine within 14 days prior to and after, or
  * any live vaccine, other than rotavirus vaccine, within 28 days prior to and after
* Previous receipt of an investigational RSV vaccine or receiving any anti-RSV product (such as ribavirin or RSV Immunoglobulin (IG) or RSV monoclonal antibody) at the time of enrollment.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of intranasal and intra-ocular medications within 3 days prior to study enrollment
* Receipt at the time of enrollment or previous receipt of salicylate (aspirin) or salicylate-containing products
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Deprived of freedom in an emergency setting, or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (6):
- United States (2):
  - Meridian Clinical Research Norfolk Site Number : 8400003, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha Site Number : 8400001, Omaha, Nebraska
- Puerto Rico (4):
  - Investigational Site Number : 6300004, Bayamón
  - Investigational Site Number : 6300002, Carolina
  - Investigational Site Number : 6300003, Guayama
  - Investigational Site Number : 6300001, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 sites in Puerto Rico from 06-Feb-2023 to 27-Dec-2024.
Pre-assignment Details: A total of 80 healthy infants/toddlers 6 to <24 months of age were randomized in contact groups of 2-3 in a 1:1 ratio to receive 2 administrations 56 days apart of either live-attenuated respiratory syncytial virus delta (Δ) non-structural (NS)2/Δ1313/I1314L vaccine (RSVt vaccine) or placebo.
Groups:
- RSVt: Participants received RSVt vaccine 0.2 milliliter (mL) as intranasal administration on Days 1 and 57
- Placebo: Participants received placebo 0.2 mL as intranasal administration in contact groups with RSVt vaccine recipients on Days 1 and 57
Period: Overall Study
Arm/Group | RSVt | Placebo
Started | 40 | 40
Completed | 35 | 38
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: Randomized set included those pediatric participants for whom a study vaccine group was allocated.
Groups:
- Placebo: Participants received placebo 0.2 milliliter (mL) as intranasal administration in contact groups with RSVt vaccine recipients on Days 1 and 57
- Total: Total of all reporting groups
Arm/Group | RSVt | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 40 | 80
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.1 (5.55) | 15.8 (5.81) | 15.4 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 24 | 17 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 29 | 27 | 56
  More than one race | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Placebo Receiving Pediatric Participants With Vaccine Virus Detected in Nasal Swabs After the First Vaccination
Description: Nasal swabs were collected to assess the presence of vaccine virus after first vaccination. Vaccine virus transmission was defined as presence of detected vaccine virus confirmed by RSVt quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay (vaccine virus shedding >=lower limit of detection [LOD=2.80 log10 copies/mL]) in pediatric participants receiving placebo. Percentages are rounded off to the tenth decimal place.
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 4, 8, 11, 15, 18 and 22
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration. Only those participants with data collected at specified timepoints are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo
Number analyzed (Participants) | 36
percentage of participants
  Day 1 | 0 [0 to 10.9]
  Day 4 | 0 [0 to 9.7]
  Day 8 | 0 [0 to 9.7]
  Day 11 | 0 [0 to 9.7]
  Day 15: number analyzed (Participants) | 35
  Day 15 | 0 [0 to 10.0]
  Day 18 | 0 [0 to 9.7]
  Day 22: number analyzed (Participants) | 34
  Day 22 | 0 [0 to 10.3]

2. Primary Outcome: Titer of Vaccine Virus Shedding in All Pediatric Participants Detected in Nasal Swabs
Description: Nasal swabs were collected to assess the shedding of the attenuated RSV vaccine strain and quantified by RSVt qRT PCR assay. Quantified virus shedding was defined as vaccine virus shedding >=lower limit of quantification (LLOQ=3.37 log10 copies/mL).
Time Frame: Pre-vaccination on Day 1 and post-vaccination on Days 4, 8, 11, 15, 18, 22, 64 and 71
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration. Only participants with quantified virus shedding at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 7 | 0
log10 copies/mL
  Day 1: number analyzed (Participants) | 0 | 0
  Day 4: number analyzed (Participants) | 0 | 0
  Day 8 | 4.33 (0.649) |
  Day 11 | 4.33 (0.617) |
  Day 15: number analyzed (Participants) | 0 | 0
  Day 18: number analyzed (Participants) | 0 | 0
  Day 22: number analyzed (Participants) | 1 | 0
  Day 22 | 4.72 |
  Day 64: number analyzed (Participants) | 2 | 0
  Day 64 | 3.55 (0.014) |
  Day 71: number analyzed (Participants) | 0 | 0

3. Primary Outcome: Percentage of Placebo Receiving Pediatric Participants With Detected Shedding Who Showed Any Genetic Sequence Variation After Each Vaccination
Description: Nasal swabs were collected to identify the difference in genetic sequence of mutated vaccine virus segments compared to the reference strain vaccine virus isolates in the vaccine virus positive swabs from pediatric participants receiving placebo after each vaccination. Detected virus shedding was defined as vaccine virus shedding >=LOD (2.80 log10 copies/mL).
Time Frame: Up to 21 days after each vaccination (Day 1 to Day 22 and Day 57 to Day 78)
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration. Only participants with detected virus shedding were included in this analysis.
Arm/Group | Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Geometric Mean Titers (GMTs) of RSV A Serum Neutralizing Antibody (nAb) Titers
Description: Serum samples were collected at specified timepoints for immunogenicity assessments. RSV A serum neutralizing antibody titers were evaluated by microneutralization (MN) assay.
Time Frame: Pre-vaccination on Day 1 (first vaccination) and Day 57 (second vaccination) and up to 28 days after second vaccination, Day 85
Population: The full analysis set included a subset of randomized pediatric participants who received at least 1 study vaccine administration. Only those participants with data collected at specified timepoints are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dilution
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 38 | 38
1/dilution
  Day 1 | 53.4 [29.7 to 95.9] | 47.9 [25.2 to 90.8]
  Day 57: number analyzed (Participants) | 34 | 37
  Day 57 | 167 [95.5 to 294] | 65.3 [30.8 to 138]
  Day 85: number analyzed (Participants) | 35 | 37
  Day 85 | 219 [126 to 382] | 60.0 [26.6 to 135]

5. Secondary Outcome: Secondary: Geometric Mean Titers of RSV Serum Anti-F Immunoglobulin G (IgG) Enzyme-linked Immuno-adsorbant Assay (ELISA) Antibody
Description: Serum samples were collected at specified timepoints for immunogenicity assessments. Antibodies to RSV F antigen were measured using the anti RSV F IgG ELISA method.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Elisa Units/mL
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 38 | 38
Elisa Units/mL
  Day 1 | 92.2 [45.5 to 187] | 85.6 [39.3 to 186]
  Day 57: number analyzed (Participants) | 34 | 37
  Day 57 | 249 [130 to 475] | 115 [49.7 to 265]
  Day 85: number analyzed (Participants) | 34 | 36
  Day 85 | 383 [205 to 714] | 129 [52.6 to 317]

6. Secondary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, i.e., pre-listed in the case report form (CRF) in terms of diagnosis and onset window post-vaccination. All participants were observed for 30 minutes after each vaccination and any unsolicited AEs that occurred during that time were recorded as immediate unsolicited AEs.
Time Frame: Up to 30 minutes after each vaccination (Days 1 and 57)
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 39 | 39
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Solicited Administration Site Reactions and Systemic Reactions
Description: A solicited reaction was an expected adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF and considered as related to the study vaccine administered. An administration site reaction was an AR at and around the administration/injection site and were commonly inflammatory reactions. Solicited systemic reactions were systemic AEs and those occurring during the specified collection period were always considered related to the vaccine even if there was evidence of alternative etiology.
Time Frame: Up to 21 days after each vaccination (Day 1 to Day 22 and Day 57 to Day 78)
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 39 | 39
Participants
  Solicited administration site reaction | 30 | 32
  Solicited systemic reaction | 26 | 25

8. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant temporally associated with the use of study vaccine, whether or not considered related to the study vaccine. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions, that is, pre-listed in the CRF in terms of diagnosis and onset window post-vaccination.
Time Frame: Up to 28 days after each vaccination (Day 1 to Day 29 and Day 57 to Day 85)
Population: The safety analysis set included those pediatric participants who received at least 1 study vaccine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVt | Placebo
Number analyzed (Participants) | 39 | 39
Participants | 8 | 12

ADVERSE EVENTS:
Time Frame: From date of first vaccination (Day 1) up to 6 months after the last study vaccination, approximately 237 days
Description: Analysis was performed on the safety analysis set
Arm/Group | RSVt | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/39 | 4/39
Other Adverse Events (participants affected / at risk) | 11/39 | 14/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSVt (N=39) | Placebo (N=39)
Bronchiolitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSVt (N=39) | Placebo (N=39)
Decreased Appetite (Metabolism and nutrition disorders) | 11 (14) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT05687279/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT05687279/SAP_001.pdf